CLINICAL TRIAL: NCT02006017
Title: Do Clinicians Want Recommendations? A Randomized Trial Comparing Evidence Summaries With and Without Evidence Based Recommendations
Brief Title: Do Clinicians Want Recommendations?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13-480
Record Dates: First submitted 2013-11-19; First posted 2013-12-09 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy Individuals (Clinicians)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): We will present to participants two general clinical scenarios. The first scenario will be accompanied by an evidence summary plus a recommendation and a second scenario will be accompanied by an evidence summary alone
  Interventions: Other: Evidence summary alone plus a recommendation; Other: Evidence summary alone
- Group B (Experimental): We will present to participants two general clinical scenarios. The first scenario will be accompanied by an evidence summary alone and a second scenario will be accompanied by an evidence summary plus a recommendation
  Interventions: Other: Evidence summary alone plus a recommendation; Other: Evidence summary alone

INTERVENTIONS:
Other: Evidence summary alone plus a recommendation
Other: Evidence summary alone

SUMMARY:
The use of the best evidence available for decision-making is nowadays an undisputed goal in health care. However, this is not always achieved in the context of clinical practice. Two of the potential solutions to bridge the gap between evidence and the clinical practice are the "evidence summaries" and the "evidence based recommendations". However, it is not clear, and frequently controversial, to what extent clinicians consider helpful recommendations accompanying evidence summaries. The investigators will explore this question by conducting a study where clinicians will be randomized to receive a clinical scenario accompanied by an evidence summary plus a recommendation and a second clinical scenario accompanied by only for an evidence summary (group A) or vice versa (Group B). The outcome will be clinicians' preferences.

ELIGIBILITY:
Inclusion Criteria:

* Were trained as Medical Doctors
* Practice primary care or general internal medicine.

Exclusion Criteria: none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2013-09-30; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Preferences | Immediately after the intervention (Survey)
  Preference: for the evidence summary plus the accompanying recommendation or for the evidence summary alone. We will assess this outcome with a 7-point Lickert scale This outcome will be assessed after the presentation of the two clinical scenarios.

SECONDARY OUTCOMES:
Understanding | Immediately after the intervention (Survey)
  Understanding: Percentage of correct answers regarding the understanding of the evidence: understanding of baseline risk, risk difference, confidence interval and quality of the evidence assessment.
Interpretation of benefits and harms | Immediately after the intervention (Survey)
  Interpretation of benefits and harms: Distribution of the interpretation of the magnitude of the benefits in comparison with harms
Intended course of action | Immediately after the intervention (Survey)
  Intended course of action: For the clinical questions related with strong recommendations, we will compare the percentage of appropriate decisions (i.e. decisions that match the strong recommendation).

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schunemann, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Neumann I, Alonso-Coello P, Vandvik PO, Agoritsas T, Mas G, Akl EA, Brignardello-Petersen R, Emparanza J, McCullagh L, De Sitio C, McGinn T, Almodaimegh H, Almodaimegh K, Rivera S, Rojas L, Stirnemann J, Irani J, Hlais S, Mustafa R, Bdair F, Aly A, Kristiansen A, Izcovich A, Ramirez A, Brozek J, Guyatt G, Schunemann HJ. Do clinicians want recommendations? A multicenter study comparing evidence summaries with and without GRADE recommendations. J Clin Epidemiol. 2018 Jul;99:33-40. doi: 10.1016/j.jclinepi.2018.02.026. Epub 2018 Mar 9. PMID 29530644